CLINICAL TRIAL: NCT04495881
Title: Effectiveness of Sitagliptin for the Treatment of Newly Diagnosed Type 2 Diabetes
Brief Title: Sitagliptin for the Treatment of Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Professor and Director, Department of Endocrinology, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-DM-Sitagliptin
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sitagliptin (Experimental): sitagliptin 100mg
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin 100mg Qd

SUMMARY:
Patients newly diagnosed with T2D will be recruited and will receive sitagliptin treatment for 3 months. The gut microbiome of the participants before and after the treatment and the effectiveness of sitagliptin treatment on type 2 diabetes will be evaluated.

DETAILED DESCRIPTION:
The dipeptidyl peptidase-4 inhibitor sitagliptin is a classic anti-diabetic drug(1) and is widely applied to both scientific research and clinical trial(2-6). This clinical trial aims to study the effectiveness of sitagliptin treatment in T2D patients and related change of gut microbiome. 50 Patients newly diagnosed with T2D will be recruited. With patient's informed consent, patient-related vital signs (such as age, height, weight, body mass index), laboratory indicators (including glycated hemoglobin, glycated albumin, low-density lipoprotein, total cholesterol, triglycerides), fasting blood glucose, insulin levels and Insulin resistance index (HOMA-IR)(7) will be recorded and analyzed. The feces of the patients will be collected to analyze the gut microbiome. All of the patients will receive the sitagliptin treatment for 3 months. The gut microbiome of the patients and the effectiveness of sitagliptin treatment on diabetes will be evaluated at indicated times during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-65 years old newly diagnosed with type 2 diabetes
* HbA1c ≥ 7%

Exclusion Criteria:

* The positive of diabetes antibodies
* Anti-diabetic drugs therapy before participation
* Pancreatitis
* Coronary artery disease
* Liver function impairment
* Renal function impairment
* History of intestinal surgery
* Chronic hypoxic diseases (emphysema and cor pulmonale)
* Infectious disease
* Hematological disease
* Systemic inflammatory disease
* Cancer
* Pregnant
* Ingesting agents known to influence glucose or lipid metabolism;
* Any antibiotics or probiotics in the past three months prior to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c change | Changes in HbA1c from baseline at 1 month and 3 months during follow-up
  Changes in HbA1c from baseline at 1 month and 3 months during follow-up

SECONDARY OUTCOMES:
fasting blood glucose change | Changes in fasting blood glucose from baseline at 1 month and 3 months during follow-up
  Changes in fasting blood glucose from baseline at 1 month and 3 months during follow-up
HOMA-IR change | Changes in HOMA-IR from baseline at 1 month and 3 months during follow-up
  Changes in HOMA-IR from baseline at 1 month and 3 months during follow-up
Glycated Albumin（GSA）change | Changes in Glycated Albumin from baseline at 1 month and 3 months during follow-up
  Changes in Glycated Albumin from baseline at 1 month and 3 months during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Q, An Y, Zhang L, Zhang Y, Wang G, Liu J. Regulation of Adropin by Sitagliptin monotherapy in participants with newly diagnosed type 2 Diabetes. BMC Endocr Disord. 2022 Dec 7;22(1):306. doi: 10.1186/s12902-022-01233-x. PMID 36476135
- [Derived] Wang Q, Ma L, Zhang Y, Zhang L, An Y, Liu J, Wang G. Effect of Sitagliptin on Serum Irisin Levels in Patients with Newly Diagnosed Type 2 Diabetes Mellitus. Diabetes Ther. 2021 Apr;12(4):1029-1039. doi: 10.1007/s13300-021-01023-z. Epub 2021 Feb 24. PMID 33625721